CLINICAL TRIAL: NCT05486156
Title: Evaluation of the Effectiveness of a Multicomponent Nature-based Intervention for Well-being and Relationship With Nature in Different Natural Areas: a Randomized Clinical Trial
Brief Title: Evaluation of a Multicomponent Nature-based Intervention for Well-being and Relationship With Nature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação Grupo Boticário de Proteção à Natureza (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A time with e-Nature
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-08

CONDITIONS: Well-being; Happiness
Keywords: Nature exposure; Multicomponent treatment; Randomized clinical trial; Well-being; Connection with nature

STUDY DESIGN:
Intervention Model Description: Participants will be separated into two groups during the study, the intervention group (IG) and the control group (CG).
Masking Description: In this study data analysts were blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention A Time with e-Nature Group (Multicomponent Nature-Based Intervention - MNBI) (Experimental): After signing the Free and Informed Consent Term, participants will be directed to a multicomponent intervention based on the experience of aesthetic, emotional and multisensory appreciation, knowledge, environmental education/interpretation and active involvement. At the end of the activity, the participants will fill in the post-intervention questionnaires, which will be applied immediately and 30 days after the intervention.
  Interventions: Other: A Time with e-Nature
- Control Group (Active Comparator): The group will do an activity made up of contact with nature during a light walk with attention directed to the senses (classical forest bathing). The trail will be accompanied by a guide who will not make any type of intervention other than offering the questionnaires to be filled in at the end of the activity and driving in the section foreseen for the activity.
  Interventions: Other: A Time with e-Nature

INTERVENTIONS:
Other: A Time with e-Nature — Integrated multisensory experience (aesthetic, emotional and knowledge) in two stages:
  1. Observation of nature through the senses (smell, hearing, sight, touch, taste) and the appreciative look.
  2. Observation focused on the local avifauna and flora during the trail accompanied by a research biologist from the group.

SUMMARY:
Randomized clinical trial to evaluate the efficacy of a multi-component nature-based intervention on clinical outcomes for visitors from different natural areas in Brazil.

DETAILED DESCRIPTION:
There is a growing scientific literature that indicates a series of benefits of contact/connection with nature for health and well-being, such as the mental health improvement, hypertension improvement, restoration of attention and memory and immune system improvement. It is already known, among other findings, that contact with nature, even indirectly, through videos and photos, can promote a greater sense of relaxation, decrease stress levels and can promote positive emotions. The adoption of nature-based interventions has been expanded, both for the prevention of chronic health conditions and the promotion of general well-being, as well as for the treatment of physical, mental and social health.

This clinical trial aims to assess the mean change in the World Health Organization well-being index, changes in self-perception of happiness, vitality, connection and engagement with nature in the pre-intervention, post-intervention and 30-day follow-up moments, in the control and intervention groups, in six different natural areas. In the multicomponent intervention, in addition to including walking in nature with attention to the senses, which will be carried out by the control group, the investigators associate other elements of a cognitive-behavioral nature, aiming human and non-human well-being. Therefore, in this health nature-based intervention, activities related to four types of experience are proposed (1- knowledge; 2- aesthetic/emotional; 3- integrated multisensory, 4- active experience). The study hypothesis is that Well-being, happiness and vitality outcomes will be more positive in the intervention group, and the connection with nature and engagement with conservation at 30 days post-intervention will be greater in the intervention group as well, due to adherence to nature-related activities that will be monitored and knowledge offered

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation;
* Signed in the Informed Consent Form (able to understand and agree to participate in the study)
* Have conditions of digital access to the link of the study questionnaires, which will be provided by the team.

Exclusion Criteria:

* Display walking difficulties;
* Participants with phobia related to elements of nature;
* History of allergies when in contact with nature.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline Well-Being Index at 30 days follow-up. | immediately pre and immediately post intervention and within 4 weeks post intervention
  The World Health Organization-5 Well-Being Index is a brief scale, composed of five questions in which the participants indicate in each one of them, based on the last two weeks, the frequency of their sensations, being 0 (at no time) and 5 (all of the time). The result is given as the sum of the numbers of each statement, with values ranging from 0, which represents the worst possible quality of life and 25, which is associated with the best possible quality of life.

SECONDARY OUTCOMES:
Change from baseline self-perception of happiness at immediate post-intervention and 30 days follow-up. | immediately pre and immediately post intervention and within 4 weeks post intervention
  A single question about ): "generally feel happy?" with an 11-point response scale (0-10) for providing a reliable and valid measure of well-being for community surveys. It is a numerical scale that varies from and used in various research ranging from 0 (extremely unhappy) to 10 (extremely happy). There is no founder of this scale being used freely as a numerical scale for several variables in which the individual can quantify in some way what is being studied. The score ranges from 0 to 10. The higher the score, the greater the happiness.
Change from baseline vitality at immediate post-intervention and 30 days follow-up. | immediately pre and immediately post intervention and within 4 weeks post intervention
  Subjective Vitality Scale consists of seven items answered on a seven-point scale, ranging from 1 (not at all true) to 7 (completely true). The respondent needs to indicate how true what the item expresses about how he is currently feeling is true.The participant needs to indicate how true what the item expresses about how they are currently feeling is true. The score ranges from 7 to 49. The higher the score, the greater vitality.
Change of Connection with Nature from baseline to 30 days post-intervention | Immediately Pre intervention and within 4 weeks post intervention
  The Nature Connection Scale (NCS) is used to verify the affective aspect of the person-environment relationship. It is composed of 14 items that are answered on a Likert Scale of points, ranging from 1 (I totally disagree) to 5 (I totally agree). The score ranges from 14 to 70. The higher the score, the greater the connection with nature.
Change from baseline nature engagement at 30 days after intervention | Immediately Pre intervention and within 4 weeks post intervention
  Nature engagement questions was developed by the project researchers themselves, with variables that trace the main motivations of the participants to go to nature, as well as variables related to the population's engagement with nature.
  In this way, it will be used to assess the frequency, motivation and access to natural areas, as well as the engagement of participants in three dimensions (values, actions taken at home in favor of nature and nature conservation actions).These questions allow to calculate the percentage of engagement for each type of action.The higher the percentage, the higher the engagement.

OTHER OUTCOMES:
Perception at the end of nature-based experience | Immediately Post intervention
  The participants emit the perception of the experience in a single word.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Roberta M Savieto, MNP, Study Chair — Hospital Israelita Albert Einstein; Denise TN Maki, MD, Study Chair — Hospital Israelita Albert Einstein; Letícia B Oliveira, BSN, Study Chair — Hospital Israelita Albert Einstein; Luccas GR Longo, MSc, Study Chair — São Paulo Municipal Secretary of Green and the Environment; Luciano M Lima, MSc, Study Chair — Butantan Institute; Erika Hingst-Zaher, Phd, Study Chair — Butantan Institute; Karina P Patricio, PhD, Study Chair — The Medical School (FMB) of São Paulo State University (Unesp),; Gustavo Borba, PhD, Study Chair — The Federal University of Technology - Paraná; Lital Bass, BSN, Study Chair — Hospital Israelita Albert Einstein; Sabrina Bomfim, Study Chair — Hospital Israelita Albert Einstein; Floriana Bertini, MD, Study Chair — Hospital Israelita Albert Einstein
Locations (6):
- Brazil (6):
  - Reserva Particular de Patrimônio Natural Salto Morato, Guaraqueçaba, Paraná
  - Parque das Neblinas, Bertioga, São Paulo
  - Parque Natural Municipal Varginha, São Paulo, São Paulo
  - Instituto Butantan, São Paulo, São Paulo
  - Parque Natural Municipal Fazenda do Carmo, São Paulo, São Paulo
  - Parque Estadual da Cantareira, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leao ER, Savieto RM, Borba GB, da Silva Victor E, Bomfim SB, Hingst-Zaher E, Lima LM, Longo LGR, de Oliveira LB, Noguchi DT, Oliveira LPG, Moredo RF, Santos CO, Menini A, Bass LM, Patricio KP, Catissi G, Rosa JM, Soldado EBR, Bertini F, de Barros CG, Kiriyama EJ. Efficacy of a multicomponent nature-based intervention on well-being and environmental engagement: A randomized clinical trial. Environ Int. 2025 Feb;196:109286. doi: 10.1016/j.envint.2025.109286. Epub 2025 Jan 19. PMID 39874898
- See also: The website features a biography and all the projects of Richard Louv, who is a writer and journalist whose published books have helped launch an international movement to connect children, families and communities to nature. — http://richardlouv.com/
- See also: Proposal of the Nature Connectedness Research Group, by University of Derby that inspired the project, based on interventions that aim to improve the relationship between the well-being of man and nature. — https://www.derby.ac.uk/research/centres-groups/nature-connectedness-research-group/
- See also: Proposal that inspired the project, based on how the natural environment can improve the health and well-being of a city's residents. With this, it is possible to bring the public of cities closer to the promotion of their well-being and nature. — https://iwun.sites.sheffield.ac.uk/
- See also: Model of nature-based health interventions as a complex adaptive system adopted in experimental group (MNBI) — https://www.frontiersin.org/journals/psychology/articles/10.3389/fpsyg.2023.1226197/full

DOCUMENTS (1):
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/56/NCT05486156/ICF_000.pdf